CLINICAL TRIAL: NCT02758678
Title: Analysis of P-selectin Expression on Platelets of Blood Between Serum Samples From Lung Cancer and Healthy Individuals by Using Raman Spectroscopy
Brief Title: Analysis of P-Selectin Expression on Platelets of Blood From Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Science and Technology Park, Center of Innovation Technologies for Human Health (Industry)
Collaborators: University in Zielona Góra (Other)
Responsible Party: Principal Investigator, Edyta Wolny-Rokicka MD.PhD, MD PhD, Science and Technology Park, Center of Innovation Technologies for Human Health
Other Study IDs: Science and Technology Park,; 2/07/2015 (Registry Identifier: bioethical commission)
Record Dates: First submitted 2016-04-18; First posted 2016-05-02 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer
Keywords: P-selectin; Lung Cancer; Raman Spectroscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A single 2 ml heparinised peripheral blood sample was centrifuges to get serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1-patients with operating tumor: 1- 23 patients with operating tumor; In 1 group the specimens of blood will be collected day before surgery and 1-2 month after surgery. Will be collected: histopathology outcomes - type carcinoma, tumore volume and before surgery: morphology and coagulation system. Will be assessed correlation between mentioned above factors and concentration of P-selectin.
  Will be compared concentration of P-selectin in 3 groups of patients.
  Serum separation and Raman spectroscopy analysis. A single 2 ml heparinised peripheral blood sample was centrifuges to get serum specimens. The Raman spectra (RS) of the solid residues from serum samples were measurement by placing 10µl of serum from the aliquots onto an aluminium substrate and allowed to dry for at least 30 min.
  Interventions: Biological: A single 2 ml heparinised peripheral blood sample
- 2-patients with advanced desease.: 2- ten patients with advanced and metastatic disease who received palliative RT (RT - radiotherapy);
  In 2 group - the specimens of blood we collected before palliative treatment-radiotherapy. Will be collected: histopathology outcomes - type carcinoma, morphology. Will be assessed correlation between mentioned factors and concentration of P-selectin. Will be compared concentration of P-selectin in 3 groups of patients. Serum separation and Raman spectroscopy analysis:
  A single 2 ml heparinised peripheral blood sample was centrifuges to get serum specimens.The Raman spectra (RS) assessed as above
  Interventions: Biological: A single 2 ml heparinised peripheral blood sample
- 3-patients with inoperable disease: In group 3 - the specimens of blood we collected before radical treatment and one month after completion treatment. Will be collected: histopathology outcomes - type carcinoma, morphology. Will be assessed correlation between mentioned above factors and concentration of P-selectin. Will be compared concentration of P-selectin in 3 groups of patients. Serum separation and Raman spectroscopy analysis:
  A single 2 ml heparinised peripheral blood sample was centrifuges to get serum specimens. The Raman spectra (RS) of the solid residues from serum samples were measurement by placing 10µl of serum from the aliquots onto an aluminium substrate and allowed to dry for at least 30 min.
  Interventions: Biological: A single 2 ml heparinised peripheral blood sample

INTERVENTIONS:
Biological: A single 2 ml heparinised peripheral blood sample — A single 2 ml heparinised peripheral blood sample was centrifuges to get serum specimens. Serum separation and Raman spectroscopy analysis:

SUMMARY:
Purpose:

Selectins are vascular cell adhesion molecules involved in adhesive interactions of leukocytes and platelets and endothelium within the blood circulation.

Plasma soluble P selectin (sP-selectin), is a one of member of selectin family, an adhesion molecule and component of the membrane of the platelet alpha granulate has been proposed as a one marker of platelet activation. In this study we evaluate of expression of P selectin on platelets of blood between serum samples from lung cancer and healthy individuals.

DETAILED DESCRIPTION:
Material and Methods:

The investigators enrolled patients with lung cancer which divided on 3 group: 1- 23 patients with operating tumor; 2-ten patients with advanced and metastatic disease who received palliative RT (RT - radiotherapy); 3-five patients with advanced inoperable disease, who received radical RT or RT + CT (CT- chemotherapy).

In 1 group the specimens of blood we collected before surgery and 1-2 month after. In 2 group - before palliative treatment and in group 3 before radical treatment and one month after completion treatment. To compare to serum specimens from patients with lung cancer was obtained plasma from healthy volunteers.

Serum separation and Raman spectroscopy analysis:

A single 2 ml heparinised peripheral blood sample was centrifuges to get serum specimens. The Raman spectra (RS) of the solid residues from serum samples were measurement by placing 10µl of serum from the aliquots onto an aluminium substrate and allowed to dry for at least 30 min. The Raman system (Renishaw inVia Microscope integrated with Leica microscope) was calibrated with a silicon standard using the Raman peak at 520 cm-1. Multiple scans were conducted on the solid residue by moving the substrate on an X - Y stage. The wavelength of excitation was 785 nm and the laser beam was focused on the surface of the sample with a 50x objective. The radius on the beam was 3.0 µm and the laser power irradiation over the sample was 5mW. Each spectrum was taken with an exposure of 30s, 10 accumulation and collected in the region from 400 to 1540 cm-1.

ELIGIBILITY:
Inclusion Criteria:

* confirmed lung cancer
* WHO 0-2
* 6 month after chemotherapy in palliative patients

Exclusion Criteria:

* double cancer
* another cancer
* chemotherapy in radical patients
* prior external beam radiation in an interview with the patient

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: both female and male participants are being studied with confirmed lung cancer
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the concentration of P-selectin in 3 groups in lung cancer patients and compared to the healthy participants. | The study started from November 2015 and will be completed in May 2016. The end of the study will be July 2016.Data will be presented up to 1 year.
  Assessment of the concentration of P-selectin in 3 groups in lung cancer patients and compare the concentration of P-selectin depends on tumor volume.Comparison between 3 groups and in the end, compared to the healthy population

CONTACTS AND LOCATIONS:
Overall Officials: Edyta I Wolny-Rokicka, MD.PhD, Study Chair — Clinicial Hospital in Zielona Góra,Radiotherapy Department ul Zyty 26, Zielona Góra, Poland
Locations (1):
- Park Naukowo-Technologiczny Uniwersytetu Zielonogórskiego Sp. z o.o., Zielona Góra, Lubusz Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
2016 - as a manuscript

REFERENCES:
- [Background] Blann AD, Lip GY. Hypothesis: is soluble P-selectin a new marker of platelet activation? Atherosclerosis. 1997 Feb 10;128(2):135-8. doi: 10.1016/s0021-9150(96)05980-1. No abstract available. PMID 9050769
- [Background] Bendas G, Borsig L. Cancer cell adhesion and metastasis: selectins, integrins, and the inhibitory potential of heparins. Int J Cell Biol. 2012;2012:676731. doi: 10.1155/2012/676731. Epub 2012 Feb 12. PMID 22505933